CLINICAL TRIAL: NCT02745613
Title: Does a Family History of Type 2 Diabetes Affect Exercise Induced Improvement in Insulin Sensitivity in a Hispanic Population?
Brief Title: Type 2 Diabetes Affect Exercise Induced Improvement in Insulin Sensitivity
Acronym: HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Sudip Bajpeyi, Associate Professor, University of Texas, El Paso
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 755513-1
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Insulin Sensitivity/Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family history of T2D (Experimental): The participants will undergo 8 weeks of combined exercise
  Interventions: Other: 8 weeks of combined exercise intervention
- No Family history of T2D (Experimental): The participants will undergo 8 weeks of combined exercise
  Interventions: Other: 8 weeks of combined exercise intervention

INTERVENTIONS:
Other: 8 weeks of combined exercise intervention — The subjects will undergo an 8 week combined exercise intervention

SUMMARY:
This study investigates weather a family history of type 2 diabetes affects exercise induced improvements in insulin sensitivity in the hispanic population

DETAILED DESCRIPTION:
A family history of T2D (FH+) is a risk factor for developing insulin resistance (which precedes T2D) and T2D (Ryder et al., 2003). Exercise training on the other hand has been shown to improve insulin sensitivity and is highly effective to prevent/manage T2D. However it is not known if early signs of insulin resistance appear before being clinically diagnosed and if the benefits of exercise which prevent/cure T2D, are limited to the offspring of Hispanic T2D parents. Therefore, the proposed study will determine 1) if normoglycemic (normal blood glucose) offspring of T2D parents are insulin resistant, using the gold standard method to measure insulin sensitivity and metabolic flexibility (ability to switch between carbohydrate and fat oxidation) 2) if 8 weeks of exercise training improves insulin sensitivity and metabolic flexibility to the same extent in FH+ compared to normoglycemic offspring of parents without any history of T2D (FH-) and 3) if 8 weeks of exercise training will change the blood, lipid and molecular profiles relevant to insulin sensitivity to same extent in FH+ compared to offspring of parents without family history of T2D (FH-).

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ Age ≤ 40 years
* 18 ≤ BMI ≤ 30 kg/m2
* Both parents are Mexican/Mexican-American)
* Sedentary lifestyle
* Less than 60 minutes/wk. of structured exercise
* Physical activity level ≤ 1.4

Exclusion Criteria:

* Evidence of significant cardiovascular disease or diabetes
* A fasting blood glucose ≥100 mg/dL
* Screening blood pressure >140/90
* Hyperlipidemia
* Use of drugs affecting energy metabolism or body weight
* Excess alcohol, drug abuse, and smoking
* Eating disorder or eating attitudes interfering with study
* Unwillingness to be abide by randomization

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 8 weeks

SECONDARY OUTCOMES:
Myokine concentrations | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sudip Bajpeyi, PhD., Principal Investigator — University of Texas, El Paso
Locations (1):
- University of Texas at El Paso, El Paso, Texas, United States